CLINICAL TRIAL: NCT02161783
Title: Treatment of Graft Failure After Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2013OC003; MT2013-06C (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Primary Graft Failure; Secondary Graft Failure
Keywords: Hematopoietic stem cell transplant
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment: This regimen consists of cyclophosphamide and fludarabine with low dose total body irradiation (TBI), followed by hematopoietic stem cell infusion.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Biological: Hematopoietic stem cell infusion

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2 IV over 1 hour given on days -6 through -2 of transplant.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 14.5 mg/kg IV over 1-2 hours given on days -6 and -5 from transplant. And Cyclophosphamide 50 mg/kg IV over 2 hours given on days +3 and +4 from transplant.
Radiation: Total Body Irradiation — TBI 200cGy in a single fraction on day -1 from transplant.
  Other Names: TBI
Biological: Hematopoietic stem cell infusion — Hematopoietic stem cell infusion given on day 0.
  Other Names: HSCT

SUMMARY:
This is a guideline for the treatment of graft failure after hematopoietic stem cell transplant (HSCT). This regimen, consisting of cyclophosphamide and fludarabine with low dose total body irradiation (TBI) is designed to promote donor engraftment by day 42 after initial graft failure.

The graft will consist of bone marrow or G-CSF mobilized peripheral blood from a haploidentical related donor. The source of stem cells will be determined by the transplant team based on factors such as patient's age, medical history, donor availability and will be according to the current University of Minnesota Blood and Marrow Transplantation Program selection guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary graft failure, as defined below, may receive a second transplant:

  * Primary graft failure is defined as not achieving an ANC ≥0.5x10^9/L for three consecutive days by day 35 - 42 following the first transplant.
  * Secondary graft failure is defined as achieving an ANC ≥0.5x10^9/L for three consecutive days by day 35 - 42, but subsequently drops below 0.5x10^9/L without recovery.
  * Loss of chimerism is defined as achieving an ANC ≥0.5x10^9/L for three consecutive, but with less than 10% CD15+ donor cells in the marrow or peripheral blood.
* Recipients should have acceptable organ function defined as:

  * Renal: creatinine < 2.0 (adults) and creatinine clearance > 30. For creatinine clearance < 70, consultation with a BMT pharmacist is necessary for chemotherapy dose adjustments.
  * Hepatic: bilirubin, AST/ALT, ALP < 10 x upper limit of normal
  * Cardiac: left ventricular ejection fraction > 40%

Exclusion Criteria:

* Uncontrolled infection at the time of transplant.
* Patients with Fanconi Anemia or other DNA breakage syndromes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Graft failure for
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-10-06 (Actual); Primary Completion 2032-01-24 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of donor engraftment | day 42
  Rate of sustained donor engraftment at day 42 post this transplant.

SECONDARY OUTCOMES:
Rate of treatment related mortality | day 100
  Rate of treatment related mortality (TRM) at day 100
Rate of survival | Day 100
  Rate of survival by day 100.
Rate of survival | 1 year
  Rate of survival at 1 year
Incidence of acute graft-versus-host disease | Day 100
  Incidence of acute graft-versus-host disease by day 100
Incidence of chronic graft-versus-host disease | 1 year
  Incidence of chronic graft-versus-host disease at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Troy C Lund, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States